CLINICAL TRIAL: NCT00946751
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Sandoz Inc. and UCB Pharma, Inc (Keppra) 750 mg Levetiracetam Tablets In Healthy Adults Volunteers Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Sandoz Inc. and UCB Pharma, Inc (Keppra) 750 mg Levetiracetam Tablets In Healthy Adults Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA15241
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Seizure
Keywords: Anticonvulsant
MeSH Terms: conditions — Seizures | interventions — Levetiracetam; Tablets

ARMS (2):
- 1 (Experimental): Levetiracetam Tablets, 750 mg (Sandoz Inc.)
  Interventions: Drug: Levetiracetam Tablets, 750 mg (Sandoz Inc.)
- 2 (Active Comparator): Keppra (Levetiracetam) Tablets, 750 mg (UCB Pharma, Inc)
  Interventions: Drug: Keppra (Levetiracetam) Tablets, 750 mg (UCB Pharma, Inc)

INTERVENTIONS:
Drug: Levetiracetam Tablets, 750 mg (Sandoz Inc.)
  Arms: 1
Drug: Keppra (Levetiracetam) Tablets, 750 mg (UCB Pharma, Inc)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Sandoz Inc. and UCB Pharma, Inc (Keppra) 750 mg Levetiracetam tablets in healthy adult volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — MDS Pharma Services